CLINICAL TRIAL: NCT05477004
Title: Ketamine Infusion for the Treatment Chronic Pain in Adults: a Prospective Observational Study to Characterize Predictors and Outcomes
Brief Title: Observational Study of Ketamine Infusions for the Treatment of Chronic Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Theresa Lii (Other)
Responsible Party: Sponsor-Investigator, Theresa Lii, Clinical Scholar, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 62561
Record Dates: First submitted 2022-07-21; First posted 2022-07-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
Keywords: ketamine; chronic pain; pain syndrome; neuropathic pain; complex regional pain syndrome; intractable pain
MeSH Terms: conditions — Chronic Pain; Somatoform Disorders; Neuralgia; Complex Regional Pain Syndromes; Pain, Intractable | interventions — Ketamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open label ketamine: Patients who receive a ketamine infusion for the treatment of chronic pain in the course of usual clinical care
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — A multi-day continuous ketamine infusion delivered intravenously at subanesthetic doses in a monitored setting
  Other Names: Ketalar

SUMMARY:
This observational study will collect prospectively specified data on patient characteristics and clinically relevant outcomes in patients who receive a ketamine infusion at Stanford Pain Management Center for the treatment of chronic pain, with the goal of identifying treatment responders and relationships between patient characteristics and treatment response.

DETAILED DESCRIPTION:
Ketamine is a type of anesthetic drug which has been used off-label to treat chronic pain. The effectiveness of intravenous ketamine and its duration of effect are not well-understood. There is high variability in response to ketamine, and it remains unclear which patient characteristics are associated with favorable outcomes. This observational study will collect a wide range of patient-reported outcomes via digital surveys: once at baseline before treatment, and up to 7 follow-up surveys for up to 12 months following a single ketamine infusion. Survey data will be supplemented by clinical data obtained from electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Has been seen at Stanford's Pain Management Center for a doctor's visit at least once.
* Is scheduled to undergo at least 1 ketamine infusion for the treatment of any chronic pain condition.
* Have a valid email address and consents to receiving surveys by email.
* Able to read, understand, and respond to English-language surveys on an electronic device such as a cell phone, tablet, or computer.
* Able to read, understand, and provide written, dated informed consent.

Exclusion Criteria:

* Has their ketamine infusion cancelled, which may occur before or after consenting to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population consists of adults who receive a ketamine infusion for the treatment of any chronic pain condition. All patients who are scheduled for a ketamine infusion through Stanford's Pain Management Center during this study's enrollment period are contacted for screening.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Patient Global Impression of Change (PGIC) in overall status; measured with PGIC Scale | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  The PGIC Scale is a single-question 7-point Likert scale ranging from "Very much improved" to "Very much worse."

SECONDARY OUTCOMES:
Change from baseline average pain intensity; measured with Numeric Rating Scale (NRS) | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  Participants rate their average pain intensity over the last 7 days using whole numbers on a 0-to-10 scale, with higher values indicative of more pain.

OTHER OUTCOMES:
Change from baseline opioid use; measured with 2 questions | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  Question 1: Participants are asked whether they have used any opioid medications since their last ketamine infusion (yes/no). Question 2: Participants are asked to rate how their opioid use has changed on a 4-point scale ranging from "I have not used any opioids since my last ketamine infusion" to "I am using more opioids after my last ketamine infusion."
Change from baseline pain catastrophizing score; measured with Pain Catastrophizing Scale - Short Form | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  Pain Catastrophizing Scale - Short Form is a 4-item scale with a total score ranging from 0-16, with higher scores indicative of more catastrophizing.
Change from baseline pain interference score; measured with PROMIS Pain Interference | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  PROMIS Pain Interference is a computerized adaptive test with results reported as a T-score (mean score of 50 and standard deviation of 10), with higher T-scores indicative of more pain interference.
Change from baseline physical function score; measured with PROMIS Physical Function | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  PROMIS Physical Function is a computerized adaptive test with results reported as a T-score (mean score of 50 and standard deviation of 10), with higher T-scores indicative of better physical function.
Change from baseline depression score; measured with PROMIS Depression | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  PROMIS Depression is a computerized adaptive test with results reported as a T-score (mean score of 50 and standard deviation of 10), with higher T-scores indicative of more depression.
Change from baseline anxiety score; measured with PROMIS Anxiety | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  PROMIS Anxiety is a computerized adaptive test with results reported as a T-score (mean score of 50 and standard deviation of 10), with higher T-scores indicative of more anxiety.
Change from baseline sleep disturbance score; measured with PROMIS Sleep Disturbance | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  PROMIS Sleep Disturbance is a computerized adaptive test with results reported as a T-score (mean score of 50 and standard deviation of 10), with higher T-scores indicative of more sleep disturbance.
Change from baseline global health score; measured with PROMIS Global Health | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  PROMIS Global Health is a computerized adaptive test with results reported as a T-score (mean score of 50 and standard deviation of 10), with higher T-scores indicative of better overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life.
Change from baseline body areas affected by pain; measured with CHOIR Body Map | 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months (or up to the time of their next ketamine infusion)
  CHOIR Body Map is a validated self-report body map where participants select areas of the body affected by pain, with a higher number of selected areas indicative of more widespread pain.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Lii, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the publication, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: IPD may be shared upon reasonable request to researchers who provide a methodologically sound proposal.